CLINICAL TRIAL: NCT04074889
Title: Study of the Effect of Probiotics on the Clinical Outcomes and Gut Microenvironment in Patients With Non-alcoholic Fatty Liver Disease: a Randomised Controlled Trial
Brief Title: The Effect of Probiotics on the Clinical Outcomes and Gut Microenvironment in Patients With Fatty Liver
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Collaborators: B-Crobes Laboratory Sdn. Bhd (Unknown); Fibronostics Pte. Ltd (Unknown); Ministry of Education, Malaysia (Other Government)
Responsible Party: Principal Investigator, Khairul Najmi, Principal Investigator, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FRGS/1/2018/SKK02/UKM/03/2
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Probiotics; Gut Liver Axis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients will be given Lactobacillus & Bifidobacterium containing probiotics [Lactobacillus acidophilus (107mg), Lactobacillus casei subsp (107mg), Lactobacillus lactis (107mg), Bifidobacterium bifidum (107mg), Bifidobacterium infantis (107mg) and Bifidobacterium longum (107mg], to be taken 1 sachet twice daily for 6 months.
  Interventions: Dietary Supplement: (Microbial cell preparation) Probiotics
- Group B (Placebo Comparator): Patients will be given placebo sachet (exactly the same packaging as active comparator) to be taken 1 sachet twice daily for 6 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: (Microbial cell preparation) Probiotics — Lactobacillus acidophilus (107mg), Lactobacillus casei subsp (107mg), Lactobacillus lactis (107mg), Bifidobacterium bifidum (107mg), Bifidobacterium infantis (107mg) and Bifidobacterium longum (107mg)
  Other Names: Hexbio
  Arms: Group A
Other: Placebo — Placebo sachet with no microbial cell preparation
  Arms: Group B

SUMMARY:
Fatty liver has been associated with high risk of progression to inflammation of the liver, liver cirrhosis (hardening of the liver), and eventually can lead to liver cancer. So far, the treatment for this condition involves controlling the cholesterol level in the body by practicing low fat diet and daily exercise. However, recently there has been evidence that alteration of the normal population of various types of bacteria that lives in the intestines may contributes to the development of fatty liver.

Probiotics is a dietary supplement containing live bacteria that is formulated to change the composition and population of the bacteria in the intestines. It is postulated that by taking specifically formulated probiotics, the alteration of the intestinal bacteria may lead to improvement of the fatty liver, leading to better daily liver function.

In this 6-month study, investigators would like to investigate the effectiveness of the probiotics in improving the liver function and in the treatment of the fatty liver. It will compare the fatty liver of patients who took the probiotics supplements compared to those who did not took it and see if there is any improvement.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is one of the common causes of chronic liver disease nowadays. NAFLD is considered as the hepatic manifestation of metabolic syndrome. In Malaysia, the prevalence of metabolic disorders such as diabetes mellitus, obesity and dyslipidemia are increasing with time. Despite the disease burden, treatments for NAFLD are currently limited due to the ongoing evolving theory of its pathogenesis.

One of the proposed mechanisms is via gut-liver axis (GLA), whereby the role of gut microbiota has been implicated. Two main components of GLA are gut microbiota and gut barrier. A change in gut microbiota composition will predispose to gut barrier dysfunction, which subsequently leads to bacterial by-products translocation into the portal circulation. Eventually, these by-products reach the liver and trigger the cascades of hepatic inflammation, leading to fatty liver and its disease progression.

The aim of this study is to investigate the role of probiotics in modulating the gut microenvironment - namely gut microbiota composition, gut barrier function and local gut inflammation, as well as its effect on the clinical outcomes in NAFLD patients.

Investigators propose a randomised, double-blind, placebo-controlled trial of 6-month duration. Investigators aim to recruit 48 NALFD patients, with either treated with probiotics or placebo. Small intestinal microbiota will be determined by 16S-rRNA sequencing and immunoreactivity of zona occludens-1 (tight junction protein in the gut barrier) and cytokines mRNA level will be measured. The degree of liver steatosis and stiffness will be assessed by using transient elastography and biochemical blood tests. All these variables will be determined pre- and post-intervention with probiotics/placebo.

This study will provide a valuable knowledge on the role of probiotics as the gut microenvironment modulator and strengthen the hypothesis of GLA involvement in the NAFLD development. Hence, probiotics can be strongly considered as one of the treatment options for non-alcoholic fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above 2. Diagnosis of NAFLD is confirmed by the presence of fatty liver detected by abdominal ultrasound and controlled attenuation parameter (CAP) score from FibroScan® of >263 3. Raised ALT level (above upper limit of normal): > 35IU/L for males and > 25 IU/L for females

Exclusion Criteria:

1. Evidence of other chronic liver diseases (as determined by clinical and standard investigations) - e.g. Hepatitis B, C infections, autoimmune hepatic disorders.
2. Evidence of acute disorders that affecting the liver - e.g. drug induced liver injury, non-Hepatitis B, C viral infection.
3. Biliary disease.
4. Liver cancer - primary hepatocellular carcinoma or liver metastasis.
5. Evidence of liver cirrhosis.
6. Alcohol intake > 20g/day for males and >10g/day for females.
7. Use of steatogenic medications within the past one months - e.g. systemic steroids, methotrexate.
8. History of bariatric surgery
9. Intake of antibiotics and/or probiotic and proton pump inhibitor within one month before the start of the study or during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Mean difference in hepatic steatosis score | 6-7 months post supplementation
  as measured by Controlled Attenuated Parameter score from Transient Elastography (Fibroscan)

SECONDARY OUTCOMES:
Mean difference in hepatic fibrosis score | 6-7 months post supplementation
  as measured by liver stiffness score from Transient Elastography (Fibroscan)
Mean difference in hepatic steatosis, inflammation and fibrosis scores | 6-7 months post supplementation
  as measured by 10 serum biomarkers (LiverFASt)
Microbiota composition of small intestine | 6-7 months post supplementation
  assessed by 16rRNA Amplicon Sequencing
Mean difference of immunoreactivity score of zona occludens-1 (ZO-1: indicator of intestinal permeability) and CD4+,CD8+, IL-8 (indicator of intestinal mucosal immune system). | 6-7 months post supplementation
  Immunohistochemistry
Mean difference in mRNA expression of genes related to inflammation (IL-6, TNF-alpha, IFN-gamma) | 6-7 months post supplementation
  Measured by serum qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Khairul Najmi Muhammad Nawawi, MBBCh BAO, Principal Investigator — The University of Malaysia Medical Centre, Kuala Lumpur, Malaysia
Locations (1):
- The University of Malaysia Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No